CLINICAL TRIAL: NCT00465959
Title: Safety, Tolerability, Pharmacokinetics, and Efficacy of Single Inhaled Administrations of Trospium Chloride Inhalation Powder (TrIP) in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Study of Trospium Chloride Inhalation Powder (TrIP) in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Collaborators: Alkermes, Inc. (Industry)
Responsible Party: Endo Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IP631-024
Record Dates: First submitted 2007-04-24; First posted 2007-04-27 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 400 mg TrIP (Experimental)
  Interventions: Drug: trospium chloride inhalation powder (TrIP)
- 800 mg TrIP (Experimental)
  Interventions: Drug: trospium chloride inhalation powder (TrIP)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: trospium chloride inhalation powder (TrIP)
  Arms: 400 mg TrIP; 800 mg TrIP
Drug: Placebo
  Arms: Placebo

SUMMARY:
To assess the effect of a single dose of TrIP on pulmonary function in patients with COPD

ELIGIBILITY:
Inclusion Criteria:

* Male or female COPD patients between the ages of 40 and 80 years
* Smoking history of at least 10 pack years
* Not currently using (or able to wash out of) any long acting bronchodilators

Exclusion Criteria:

* Candidate on a waiting list for surgery while on study
* Using long-term oxygen therapy
* Hospitalization for COPD exacerbation

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-04; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy (measured by spirometry) of TrIP will be assessed in patients with chronic obstructive pulmonary disease.

CONTACTS AND LOCATIONS:
Locations (1):
- United States Investigational Site, Spartanburg, South Carolina, United States